CLINICAL TRIAL: NCT03603847
Title: Prospective Study of the Prognostic Value of New Markers in Adults With ALK-positive Large Anaplastic Lymphoma
Status: Completed | Type: Observational
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other); Fondation ARC (Other); Pfizer (Industry); Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: ALK-OBS
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Positive
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, constitutional DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the prognostic value on the complete metabolic response rate (MCR), the incidence of relapse / progression, the Progression Free Survival (PFS) and the Overall Survival (OS).

* at diagnosis
* after the first cycle of CHOEP (early evaluation)
* at the end of treatment

DETAILED DESCRIPTION:
ALK-positive anaplastic large cell (anaplastic large-cell lymphoma, ALCL) is a rare adult disease for which almost all published studies are retrospective. The overall survival (OS) at 5 years varies from 70 to 87%. A recent international pooled analysis showed that the International Prognostic Index (IPI) had good predictive value for the PFS and the OS.

In children, new prognostic factors have been identified: the titre of circulating anti-ALK antibodies (inverse correlation between the antibody titre and the prognosis), the detection of a NPM-ALK transcript in the blood at diagnosis (minimal disseminated disease, MDD); correlation between MDD positivity and pejorative prognosis) and its minimal residual disease (MRD), and the histological subtype (common versus small cells / lymphohistiocytic).

The predictive value of the oncogenic profile of ALK-positive ALCL and circulating tumor DNA will be studied in this study.

* At diagnosis (before starting treatment):
* Cycle 2 Day 1 (before starting cycle 2 treatment):
* At the end of treatment evaluation:

  40 patients treated with 6 cycles of CHOEP every 3 weeks and 1 lumbar puncture at diagnosis with intrathecal prophylaxis with methotrexate will be included prospectively.

During a 2-year period, relapses / progressions and patient deaths will be monitored for the calculation of the incidence of relapse / progression, progression free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

Over 18 years old Diagnosed with Anaplastic large-cell lymphoma ALK+

Planned treatment : 6 cycles of CHOEP 21

Planned lumbar puncture at diagnosis or at the first cycle with intrathecal prophylaxis with methotrexate (15 mg) at the first cycle

Planned interim positron emission tomograph (PET)-scan after 3 cycles of treatment and at the end of treatment according to the center standard of care

Exclusion Criteria:

Involvement of the central nervous system

Intent of Autologous stem-cell transplant in first line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Anaplastic large-cell lymphoma ALK+
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Prognostic value of biological parameters on the complete metabolic response rate (MCR) | Day 0

SECONDARY OUTCOMES:
Prognostic value of biological parameters on the complete metabolic response rate (MCR) | 1 month
Prognostic value of biological parameters on the complete metabolic response rate (MCR) | 2 years
Prognostic value of biological parameters on the incidence of relapse | Day 0
Prognostic value of biological parameters on the incidence of relapse | 1 month
Prognostic value of biological parameters on the incidence relapse | 2 years
Prognostic value of biological parameters on the Progression Free Survival (PFS) | Day 0
Prognostic value of biological parameters on the Progression Free Survival (PFS) | 1 month
Prognostic value of biological parameters on the Progression Free Survival (PFS) | 2 years
Prognostic value of biological parameters on the Overall Survival (OS) | Day 0
Prognostic value of biological parameters on the Overall Survival (OS) | 1 month
Prognostic value of biological parameters on the Overall Survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David SIBON, MD, Principal Investigator — Hôpital Necker-Enfants Malades
Locations (15):
- France (15):
  - CHU Amiens - Hôpital Sud, Amiens
  - CHU d'Estaing, Clermont-Ferrand
  - APHP - Hopital Henri Mondor, Créteil
  - CHU Grenoble, Grenoble
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - Institut Paoli Calmette, Marseille
  - APHP - Hôpital Necker, Paris
  - APHP - Hôpital Saint Louis, Paris
  - CHU Bordeaux - Centre François Magendie, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rennes - Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CHRU de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sibon D, Fournier M, Briere J, Lamant L, Haioun C, Coiffier B, Bologna S, Morel P, Gabarre J, Hermine O, Sonet A, Gisselbrecht C, Delsol G, Gaulard P, Tilly H. Long-term outcome of adults with systemic anaplastic large-cell lymphoma treated within the Groupe d'Etude des Lymphomes de l'Adulte trials. J Clin Oncol. 2012 Nov 10;30(32):3939-46. doi: 10.1200/JCO.2012.42.2345. Epub 2012 Oct 8. PMID 23045585
- [Background] Damm-Welk C, Mussolin L, Zimmermann M, Pillon M, Klapper W, Oschlies I, d'Amore ES, Reiter A, Woessmann W, Rosolen A. Early assessment of minimal residual disease identifies patients at very high relapse risk in NPM-ALK-positive anaplastic large-cell lymphoma. Blood. 2014 Jan 16;123(3):334-7. doi: 10.1182/blood-2013-09-526202. Epub 2013 Dec 2. PMID 24297868
- [Background] Damm-Welk C, Pillon M, Woessmann W, Mussolin L. Prognostic factors in paediatric anaplastic large cell lymphoma: role of ALK. Front Biosci (Schol Ed). 2015 Jun 1;7(2):205-16. doi: 10.2741/S434. PMID 25961696
- [Background] Lamant L, McCarthy K, d'Amore E, Klapper W, Nakagawa A, Fraga M, Maldyk J, Simonitsch-Klupp I, Oschlies I, Delsol G, Mauguen A, Brugieres L, Le Deley MC. Prognostic impact of morphologic and phenotypic features of childhood ALK-positive anaplastic large-cell lymphoma: results of the ALCL99 study. J Clin Oncol. 2011 Dec 10;29(35):4669-76. doi: 10.1200/JCO.2011.36.5411. Epub 2011 Nov 14. PMID 22084369